CLINICAL TRIAL: NCT06083883
Title: Phase I/Ib Study of Adoptive NK Expressing an Affinity-enhanced T-cell Receptor (TCR) Reactive Against the NY-ESO-1-specific Cord Blood-derived NK Cells (NY-ESO-1 TCR/IL-15 NK) in Conjunction With Lymphodepleting Chemotherapy for the Management of Advanced Synovial Sarcoma and Myxoid/Round Cell Liposarcoma
Brief Title: Phase I/Ib Study of NK Expressing an Affinity-enhanced T-cell Receptor (TCR) Against the NY-ESO-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0289; NCI-2023-08752 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Synovial Sarcoma; Myxoid/Round Cell Liposarcoma
MeSH Terms: conditions — Sarcoma, Synovial; Liposarcoma, Myxoid | interventions — fludarabine phosphate; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation - Inpatient and Outpatient (Experimental): Participants will be assigned to receive a dose level of NK cells based on when the participants joins the study. Up to 6 participants will be enrolled at each dose level. If no intolerable side effects are seen after the first 3-6, the next group of participants will get at higher dose. Up to 4 dose levels of NK cells will be tested. If the first dosing group shows intolerable side effects, a lower dose will be tested.
  Interventions: Drug: Fludarabine phosphate; Drug: NY-ESO-1 TCR/IL-15 NK; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Fludarabine phosphate — Given by IV (vein)
  Other Names: Fludarabine; Fludara®
Drug: NY-ESO-1 TCR/IL-15 NK — Given by IV (vein)
Drug: Cyclophosphamide — Given by IV (vein)
  Other Names: Cytoxan®; Neosar®

SUMMARY:
The goal of this clinical research study is to find a recommended dose of donated NK cells that can be given along with chemotherapy to patients with advanced cancers. The safety and effects of this therapy will also be studied.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the safety and optimal cell dose of adoptive NK expressing an affinity-enhanced Tcell receptor (TCR) reactive against the NY-ESO-1- r (NY-ESO-1 TCR/IL-15 NK) in patients with advanced synovial sarcoma and myxoid/round cell liposarcoma
2. To determine the antitumor activity of adoptive CB-specific NK cells expressing an affinityenhanced T-cell receptor (TCR) reactive against the NY-ESO-1- (NY-ESO-1 TCR/IL-15 NK).

Secondary Objectives

1. To investigate the correlation between the percentage of NY-ESO-1 in the pre-treatment sample of the tumor, and the tumor response to the treatment.

Exploratory Objectives

1. To quantify the persistence of infused allogeneic adoptive NK expressing an affinity-enhanced T-cell receptor (TCR) reactive against the NY-ESO-1-specific CB-derived NK cells (NY-ESO-1 TCR/IL15 NK) in the recipient.
2. To conduct comprehensive immune reconstitution studies.
3. To obtain preliminary data on quality of life and patient experience.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with all cancer histology, with an HLA-A*02:01, HLA-A*02:05 or HLA-A*02:06 positive and a positive expression of NY-ESO-1 (>/= 50% tumor cells 2+ or 3+ by IHC) in the preenrollment tumor sample, for the dose escalation cohort. NY-ESO expression must be confirmed at MDACC prior to study entry.
2. Patients with histologically confirmed synovial sarcoma (cohort 1) or myxoid/round cell liposarcoma (cohort 2), with an HLA-A*02:01, HLA-A*02:05 or HLA-A*02:06 positive and a positive expression of NY-ESO-1 (>/= 50% tumor cells 2+ or 3+ by IHC) in the pre-enrollment tumor sample, for the expansion cohorts. Archival samples will be permitted for screening. NY-ESO expression must be confirmed at MDACC prior to study entry.
3. Patients must meet disease-specific eligibility criteria (see below).
4. Patients must have relapsed or become refractory to standard of care treatment and must have received at least one prior line of systemic therapy including either doxorubicin and/or ifosfamide (synovial sarcoma and MRCLS) or trabectedin (MRCLS).
5. Patients must have measurable disease per the RECIST v1.1 at enrollment.
6. Patients must be at least 2 weeks from last cytotoxic chemotherapy at the time of first administration of lymphodepleting chemotherapy. Patients may continue tyrosine kinase inhibitors or other targeted therapies until at least 3 days prior to administration of lymphodepleting chemotherapy.
7. Patients must be at least 3 months from any cell therapy for malignancy.
8. Eastern Cooperative Oncology Group performance status 0-1 (Appendix A).
9. Adequate organ function at screening, as defined by the following:

   1. Renal: Serum creatinine ≤ 1.5 mg/dL or estimated glomerular filtration rate (Chronic Kidney Disease Epidemiology Collaboration equation) ≥45 ml/min/1.73 m2
   2. Hepatic: alanine transaminase (ALT)/aspartate transaminase (AST) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5 x ULN if documented liver metastases, total bilirubin ≤ 1.5 mg/dL or ≤ 3.0 mg/dL for patients with Gilbert's Syndrome. No history of liver cirrhosis and no ascites.
   3. Cardiac: Cardiac ejection fraction ≥ 50%, no clinically significant pericardial effusion as determined by echocardiogram (ECHO) or multigated acquisition (MUGA) scan, and no symptomatic cardiac disease or history of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
   4. Pulmonary: No clinically significant pleural effusion (per principal investigator [PI] judgement), and baseline oxygen saturation ≥ 92% on room air,
   5. Hematological: absolute neutrophil count (ANC) ≥ 1000/mm3, platelet count ≥ 75,000/mm3, and hemoglobin ≥ 8 g/dL
   6. Coagulation: International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 ULN. Patients on therapeutic doses of anticoagulation medication must have INR and/or aPTT ≤ the upper limit of the therapeutic range for intended use.
10. Able to provide written informed consent.
11. Aged 16-80 years.
12. Weight ≥40 kg.
13. All male and female patients who are able to have children must practice effective birth control while on study therapy and for up to 3 months post completion of study therapy. Acceptable forms of birth control for female patients include: hormonal birth control, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence. Female patients who become pregnant or suspect pregnancy must immediately notify their doctor. Females patients who become pregnant will be taken off study. Men who are able to have children must use effective birth control while on the study therapy.

    Acceptable forms of birth control for male patients include: condom with spermicide or abstinence. If the male patient fathers a child or suspects that he has fathered a child while on the study, he must immediately notify his doctor.
14. Negative serum or urine beta human chorionic gonadotropin pregnancy test for females of childbearing potential (defined as not postmenopausal for 24 months or no previous surgical sterilization or lactating females) at screening.
15. Signed consent to long-term follow-up on protocol PA17-0483.
16. Disease-specific inclusion criteria
17. Advanced solid tumors a. Patients with locally advanced and/or metastatic solid tumors may be enrolled in the dose escalation phase. Patients must have received at least one prior line of standard therapy.

18 Synovial Sarcoma (SS)

a. Patients must have a histologically confirmed diagnosis of synovial sarcoma with a confirmation by the presence of a translocation between SYT on the X chromosome and SSX1, SSX2 or, SSX4 on chromosome 18 (may be presented in the pathology report as t (X; 18)).

19. Myxoid/round cell liposarcoma (MRCLS)

a. Patients must have histologically confirmed myxoid/round cell liposarcoma with a confirmation by the presence of the reciprocal chromosomal translocation t(12;16)(q13;p11) or t(12; 22) (q13;q12).

Exclusion Criteria:

1. Presence of clinically significant ≥ Grade 2 toxicity from previous anticancer treatment, as determined by the PI.
2. Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management or not responding to appropriate therapy. Note: Patients with simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
3. Known Active hepatitis B or C.
4. Known human immunodeficiency virus with detectable viral load.
5. Presence of active neurological disorder(s).
6. Active autoimmune disease within 12 months of enrollment (excluding low-grade psoriasis or well-controlled autoimmune thyroid disease).
7. Amyloidosis or POEMS syndrome.
8. Symptomatic or uncontrolled central nervous system involvement or signs of cord compression.

   In the case radiation therapy is indicated, the washout must be at least 14 days.

   Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using corticosteroids for at least 7 days prior to trial treatment.
9. Patients must not have any other malignancies within the past 2 years except for in situ carcinoma of any site, adequately treated (without recurrence post resection or post radiotherapy) carcinoma of the cervix or basal or squamous cell carcinomas of the skin, or active non-lifethreatening second malignancy that would not, in the investigator's opinion, potentially interfere with the patient's ability to participate and/or complete this trial. Examples include but are not limited to: urothelial cancer Grade Ta or T1 and adenocarcinoma of the prostate treated by active surveillance.
10. Presence of any other serious medical condition that may endanger the patient at investigator's discretion, including but not limited to:

    * New York Heart Association Class III or IV heart failure
    * Myocardial infarction or stroke ≤ 26 weeks prior to NY-ESO-1 TCR/IL-15 NK cell infusion
    * Unstable angina within ≤ 13 weeks prior to NY-ESO-1 TCR/IL-15 NK cell infusion unless the underlying disease has been corrected by procedural intervention (e.g., stent, bypass)
    * Severe aortic stenosis.
    * Uncontrolled arrhythmia, considered per PI evaluation.
    * Congenital long QT syndrome.
    * Documentation, during the screening process, of a QTc > 470 milliseconds by Fredericia criteria (QTcF) based on the average of 3 electrocardiograms (ECGs) taken approximately 1 minute apart and all within 10 minutes of each other. The patient should be reclining for 5 minutes prior to ECGs. Local readings may be used for this exclusion criterion.
11. Major surgery < 4 weeks prior to first dose of lymphodepleting chemotherapy.
12. Concomitant use of other investigational agents.
13. Concomitant use of other anticancer agents.
14. Previously received any anti-NY-ESO-1 therapy.
15. Patients receiving systemic steroid therapy at time of enrollment, with an exception for topical, ocular, intranasal, and inhaled corticosteroids, or systemic corticosteroids at an equivalent dose ≤ 10 mg of prednisone daily (physiological substitutive doses are allowed).
16. Received antithymocyte globulin within 14 days or Campath within 28 days of enrollment.
17. Patients receiving immunosuppressive therapy.
18. Patients who received live vaccines within 30 days prior enrollment.
19. Pregnant or breastfeeding.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: John Livingston, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org